CLINICAL TRIAL: NCT07052825
Title: The Role of Capsular Tension Rings in Intraocular Lens Stability in High Myopia Cataract Patients: A Prospective Self-Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jin Yang (Other)
Responsible Party: Sponsor-Investigator, Jin Yang, Chief Physician, Eye & ENT Hospital of Fudan University
Organization: Eye & ENT Hospital of Fudan University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM CTR; 82171039 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2025-06-29; First posted 2025-07-07 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-06

CONDITIONS: High Myopia; Cataract
Keywords: Capsular Tension Ring（CTR）, High Myopia, Intraocular lens, Tilt, Decentration, Visual Quality
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This is a self-controlled study. Each participant receives cataract surgery in both eyes, with one eye randomly assigned to CTR implantation and the fellow eye without CTR. The two eyes serve as within-subject comparators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTR implantation (Experimental): Phaco+IOL with CTR implantation
  Interventions: Procedure: CTR implantation
- NCTR (No Intervention): Phaco+IOL without CTR implantation

INTERVENTIONS:
Procedure: CTR implantation — Phaco+IOL with CTR implantation
  Arms: CTR implantation

SUMMARY:
Study Purpose:

This prospective, self-controlled clinical study aims to evaluate the impact of capsular tension rings (CTR) on intraocular lens (IOL) stability in high myopia patients undergoing bilateral cataract surgery. Each patient will receive CTR implantation in one eye, with the fellow eye serving as control. Postoperative outcomes, including visual acuity, refraction, IOL positioning, and visual quality, will be compared between eyes to assess the effectiveness of CTR.

Study Methods:

Eligible participants (axial length ≥ 26.0 mm) will undergo femtosecond-assisted phacoemulsification with identical IOLs implanted in both eyes. One eye will be randomly assigned to receive a CTR. All surgeries will be performed by the same surgeon. Follow-up will be conducted at 1 day, 1 week, 1 month, 3 months, and 6 months postoperatively. Assessments will include UCVA, BCVA, refractive error, anterior segment OCT, IOL decentration and tilt, and visual quality (iTrace).

Sample Size and Population:

A total of 60 patients (120 eyes) will be enrolled. Inclusion criteria include age ≥ 18 years and bilateral cataracts with high myopia. Exclusion criteria include other ocular diseases, history of severe ocular trauma, or poor visual potential. Patients will be stratified by axial length into three groups: ≤28 mm, 28-30 mm, and >30 mm.

Study Procedure:

After informed consent and baseline examinations (including ocular biometry and imaging), patients will undergo surgery and be followed at specified intervals. All data will be managed securely. Comparative analysis between CTR and non-CTR eyes will be performed to evaluate the effect of CTR on IOL stability and visual outcomes in highly myopic cataract patients.

DETAILED DESCRIPTION:
Study Purpose:

This study aims to evaluate the effect of capsular tension rings (CTR) on intraocular lens (IOL) stability in cataract patients with high myopia. Each patient will undergo cataract surgery in both eyes, with one eye receiving a CTR and the other eye not receiving a CTR, using the same IOL model in both eyes. Postoperative visual quality and IOL stability will be compared between the two eyes. The study will analyze changes in postoperative visual acuity, refraction, ocular parameters, anterior segment morphology, and IOL positioning to assess the effect of CTR implantation on visual outcomes in highly myopic patients.

Study Methods:

This is a prospective, self-controlled clinical study involving cataract patients with high myopia (axial length ≥ 26.0 mm) scheduled for bilateral cataract surgery. Patients will undergo femtosecond-assisted phacoemulsification and IOL implantation in both eyes, with one eye randomly assigned to receive a CTR and the other not. All procedures will be performed by the same surgeon to ensure consistency. Postoperative follow-up visits will be scheduled at 1 day, 1 week, 1 month, 3 months, and 6 months. Evaluation indicators include uncorrected and best corrected visual acuity (UCVA, BCVA), refractive status, intraocular pressure, anterior segment morphology (anterior segment OCT), IOL decentration and tilt (using anterior segment images), and visual quality (iTrace).

Sample Size and Study Population:

The estimated sample size is 60 patients (i.e., 120 eyes). Each patient will receive CTR implantation in one eye and serve as their own control in the fellow eye. Inclusion criteria: age ≥ 18 years, bilateral cataracts with high myopia eligible for surgery. Exclusion criteria: ocular comorbidities (e.g., glaucoma, retinal disease), history of major ocular trauma or surgery, and other causes of vision loss. Patients will be grouped based on axial length: Group A (AL ≤ 28 mm), Group B (28 mm < AL ≤ 30 mm), and Group C (AL > 30 mm).

Study Procedure:

Participants will be recruited after signing informed consent and passing pre-screening assessments. All subjects will receive detailed explanations regarding study purpose, procedures, risks, and postoperative care. Baseline examinations will include biometry, axial length, anterior segment measurements, and corneal topography. After surgery, patients will be followed up at 1 day, 1 week, 1 month, 3 months, and 6 months. Examinations include visual acuity, refraction, intraocular pressure, IOL position (decentration and tilt via anterior segment OCT), and visual quality analysis (iTrace). All data will be securely managed, and the final analysis will compare visual outcomes and IOL stability between the CTR and non-CTR eyes in highly myopic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosed with bilateral age-related cataracts and scheduled for phacoemulsification with IOL implantation in both eyes.
3. High myopia in both eyes, defined as axial length (AL) ≥ 26.0 mm.
4. No significant difference in axial length between the two eyes (e.g., interocular AL difference < 1.0 mm).
5. Willingness and ability to undergo bilateral surgery within a short interval (e.g., within 1-2 weeks).
6. Able to provide informed consent and comply with the study protocol and follow-up visits.

Exclusion Criteria:

1. History of ocular trauma, surgery, or intraocular inflammation in either eye.
2. Presence of other ocular diseases that may affect visual outcomes, such as glaucoma, diabetic retinopathy, macular degeneration, or corneal opacity.
3. Evidence of zonular weakness, pseudoexfoliation, or significant phacodonesis preoperatively.
4. Severe dry eye or poor fixation that may interfere with postoperative imaging.
5. Systemic diseases affecting visual function (e.g., uncontrolled diabetes, neurologic disorders).
6. Participation in other clinical trials that may affect the study outcomes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Tilt and Decentration | Postoperative follow-up visits will be scheduled at 1 day, 1 week, 1 month, 3 months, and 6 months
  measured by using anterior segment OCT

SECONDARY OUTCOMES:
Anterior Capsular Contraction | 1 day, 1 week, 1 month, 3 months, and 6 months postoperatively
  Measured by Anterior Segment Photography and ImageJ
visual acuity | 1 day, 1 week, 1 month, 3 months, and 6 months postoperatively
  UDVA AND BCVA
Visual Quality | 1 day, 1 week, 1 month, 3 months, and 6 months postoperatively
  Measured by iTace

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yang, Study Chair — Fudan University
Locations (1):
- Eye and ENT hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No